CLINICAL TRIAL: NCT04576819
Title: Role and Mechanisms of Lipid and Lipoprotein Dysregulation in Sepsis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201903081-N; 1R01GM133815-01A1 (NIH)
Record Dates: First submitted 2020-09-25; First posted 2020-10-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Sepsis; Shock, Septic
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection for serum, plasma, leukocytes samples for RNA extraction, and PBMC collection for RNA sequence analysis. DNA samples may also be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis cohort: Inclusion criteria
  * Patients meeting the Sepsis-3 definition of sepsis or septic shock (the sequential organ failure assessment (SOFA) score will be used for organ failure assessment for Sepsis-3 criteria)
  * Treatment with an institutional, evidence-based guideline management bundle for sepsis
  * Within 24 hrs of sepsis recognition
  Exclusion criteria:
  * alternative/confounding diagnosis causing shock (e.g., myocardial infarction or pulmonary embolus),
  * uncontrollable source of sepsis (e.g., irreversible disease state such as unresectable dead bowel),
  * advanced directives limiting resuscitative efforts,
  * organ transplant recipient on immunosuppressive agents,
  * known pregnancy,
  * inability to obtain informed consent,
  * HIV/AIDS with CD4 count < 200,
  * absolute neutrophil count < 500

SUMMARY:
Lipids and lipoproteins (cholesterol and lipid metabolites) are present in sepsis and are highly biologically active regulators of inflammation, but currently the changes in lipid and lipoprotein homeostasis during sepsis are not well understood. This project will investigate the changes in lipid and lipoprotein function, oxidation, metabolites, and changes in gene expression to further our understanding of dysregulated lipid and lipoprotein metabolism in sepsis. We will analyze a bank of samples and make associations with important clinical outcomes (early death, chronic critical illness and sepsis recidivism) as supported by our published work, and will confirm our findings in a small prospective cohort of sepsis patients.

DETAILED DESCRIPTION:
This study will use biobanked samples from a diverse cohort of 165 sepsis patients (UF Jacksonville and UF Gainesville) and will confirm findings in a small prospective cohort of 50 patients. The following will be tested in patient samples:

Aim 1: Test and compare HDL and LDL function (oxidation/transport) in sepsis patients by clinical outcomes of rapid recovery, early death, CCI, and sepsis recidivism.

Aim 2: Determine the changes in lipid homeostasis and patterns of inflammation that occur in sepsis patients by outcome.

Aim 3: Characterize cholesterol & lipoprotein-specific metabolic gene expression in whole blood leukocytes and peripheral blood mononuclear cells from sepsis patients.

ELIGIBILITY:
Inclusion criteria:

* Patients meeting the Sepsis-3 definition of sepsis or septic shock
* Treatment with an institutional, evidence-based guideline management bundle for sepsis within 24 hrs of sepsis recognition
* Sequential organ failure assessment (SOFA) score will be used for organ failure assessment.

Exclusion criteria:

* a) alternative/confounding diagnosis causing shock (e.g., myocardial infarction or pulmonary embolus)
* b) uncontrollable source of sepsis (e.g., irreversible disease state such as unresectable dead bowel)
* c) advanced directives limiting resuscitative efforts
* d) organ transplant recipient on immunosuppressive agents
* e) known pregnancy
* f) inability to obtain informed consent
* g) HIV/AIDS with CD4 count < 200, h) absolute neutrophil count < 500. These criteria are justified by numerous prior studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients meeting the Sepsis-3 definition of sepsis and being treated with institutional evidence-based care bundles.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Chronic Critical Illness or Early Death | 14 days from sepsis onset
  CCI defined as admission to ICU > 14 days total with organ dysfunction, Early death defined as death within 14 days of hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Faheem Guirgis, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Augustin B, Wu D, Black LP, Bertrand A, Sulaiman D, Hopson C, Jacob V, Shavit JA, Hofmaenner DA, Labilloy G, Smith L, Cagmat E, Graim K, Datta S, Reddy ST, Guirgis FW. Multiomic molecular patterns of lipid dysregulation in a subphenotype of sepsis with higher shock incidence and mortality. Crit Care. 2024 Dec 24;28(1):431. doi: 10.1186/s13054-024-05216-3. PMID 39716214